CLINICAL TRIAL: NCT06057779
Title: The Effect of Loading Speed and Intensity During Exercise on the Immediate Changes in Achilles Tendon Thickness and Stiffness: a Randomised Crossover Trial
Brief Title: The Effect of Loading Speed and Intensity During Exercise on the Immediate Structural Changes in the Achilles Tendon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ONZ-2023-0238
Record Dates: First submitted 2023-08-23; First posted 2023-09-28 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Achilles Tendinopathy
Keywords: Achilles tendon

STUDY DESIGN:
Intervention Model Description: Repeated measure design
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor was blinded to the specific intervention (protocol type); due to the nature of the interventions, participants were aware of the exercise intervention they were performing each week. However, participants will not be informed of the hypothesis of the study nor will this be disclosed at any time in written materials or verbal interactions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Slow and heavy exercise therapy (Other): Participants perform eccentric heel drop exercises into maximal dorsiflexion at slow speed.
  Interventions: Other: Slow and heavy exercise therapy
- Slow and light exercise therapy (Other): Participants perform eccentric heel drop exercises into neutral ankle position at slow speed.
  Interventions: Other: Slow and light exercise therapy
- Fast and heavy exercise therapy (Other): Participants perform eccentric heel drop exercises into maximal dorsiflexion at fast speed.
  Interventions: Other: Fast and heavy exercise therapy

INTERVENTIONS:
Other: Slow and heavy exercise therapy — 6 sets of 10 single leg isolated eccentric heel drops into maximal dorsiflexion at an exercise speed of 0.33 Hz, with 1-min rest period between each set.
  Arms: Slow and heavy exercise therapy
Other: Slow and light exercise therapy — 6 sets of 10 single leg isolated eccentric heel drops into neutral ankle position at an exercise speed of 0.33 Hz, with 1-min rest period between each set.
  Arms: Slow and light exercise therapy
Other: Fast and heavy exercise therapy — 6 sets of 30 single leg isolated eccentric heel drops into maximal dorsiflexion at an exercise speed of 1 Hz, with 1-min rest period between each set.
  Arms: Fast and heavy exercise therapy

SUMMARY:
Aim: To assess the influence of loading speed and intensity during eccentric heel drop exercise on the immediate changes in Achilles tendon thickness and stiffness in healthy controls.

Intervention: Three eccentric heel drop exercise protocols, different in loading speed and/or loading intensity will be compared. Each participant will perform a single protocol per session in a random sequence at 1-week intervals.

Participants: a total of 34 healthy athletes will be included.

Outcome measure: tendon thickness and stiffness will be measured at baseline and immediately following intervention with ultrasound imaging (B-mode) and shear wave elastography, respectively.

Discussion: the study will determine whether an eccentric exercise intervention involving a low loading speed and high intensity could maximize the immediate reduction in thickness and associated increase in stiffness of the Achilles tendon compared with interventions involving a higher loading speed and lower intensity.

DETAILED DESCRIPTION:
Mechanical loading of the Achilles tendon during isolated eccentric contractions induces immediate changes in its structural properties. However, it is not known whether the loading speed and intensity has any impact on these changes. Therefore, this study aims to investigate the influence of loading speed and intensity during eccentric heel drop exercises on the immediate changes in Achilles tendon thickness and stiffness in healthy controls.

Each participant will perform eccentric heel-drops on their dominant leg with and a fully extended knee, and with additional 20% body weight (added via a weighted backpack). Participants will stand with the forefoot of the tested limb on the edge of a step, with the ankle maximally plantar flexed and with body weight centred on this limb. Eccentric loading occurs when the participant lowers the heel to a predetermined angle and speed (depending on the type of intensity and speed cfr infra). In order to return to baseline, the body mass will therefore be shifted to the non-dominant leg to raise the body. Visual feedback (monitor) will be in front of the subjects and the exercise parameters (velocity and ankle angle) will be guided by software guidelines (Ultium Motion).

Three protocols will be compared that differ in execution speed (namely a fast protocol; 1 Hz: 1 second per repetition versus a slow protocol; 0.33 Hz: 3 seconds per repetition) and loading intensity (namely heavy; exercise into maximal dorsiflexion versus light; exercise into neutral ankle position).

Protocol 1 (=Heavy x Slow): subjects perform eccentric heel drops from a maximal plantarflexion position to a maximal dorsiflexion position at a speed of 0.33 Hz, i.e. 3 seconds per movement cycle.

Protocol 2 (=Heavy x Fast): subjects perform eccentric heel drops from a maximal plantarflexion position to a maximal dorsiflexion position at a speed of 3 Hz, i.e. 1 seconds per movement cycle.

Protocol 3 (=Light x Slow): subjects perform eccentric heel drops from a maximal plantarflexion position to a neutral ankle position at a speed of 0.33 Hz, i.e. 3 seconds per movement cycle.

Participants will perform one exercise protocol per session, in a random order, and the interval between each session is one week. Six sets will be performed per session, with one minute of rest between each set. In order to ensure that the Achilles tendon's time under tension is the same for each protocol (180 seconds), 30 repetitions will performed per set for the fast protocol and 10 repetitions for the slow protocol. The approximate duration of each intervention will be 15 minutes. Before and immediately after each protocol, the structural properties of the Achilles tendon, 20 mm proximal to the calcaneal posterosuperior border, will be assessed. These properties include tendon thickness (anteroposterior diameter (mm), cross-sectional arae (mm2)), and tendon stiffness by shear wave elastography (m/s).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 55 years
* Participate in recreational or competitive sport (at least 1x/week)

Exclusion Criteria:

* History of Achilles tendinopathy
* Presence of rheumatological disease
* Not able to complete an exercise programme

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Achilles tendon thickness | Baseline and immediately following each protocol
  Tendon anteroposterior diameter will be assessed 20 mm proximal to the posterosuperior calcaneal border using ultrasound imaging. The Achilles tendon is scanned at rest with the subject in the prone position and the foot passively maintained in a neutral position.
Achilles tendon cross-sectional area | Baseline and immediately following each protocol
  Tendon cross-sectional area of the Achilles tendon will be assessed 20 mm proximal to the posterosuperior calcaneal border using ultrasound imaging. The Achilles tendon is scanned at rest with the subject in the prone position and the foot passively maintained in a neutral position.
Achilles tendon stiffness | Baseline and immediately following each protocol
  Echogenicity of the Achilles tendon will be assessed 20 mm proximal to the posterosuperior calcaneal border using shear wave elastography. The Achilles tendon is scanned at rest with the subject in the prone position and the foot passively maintained in a 30° plantar flexion.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Vanden Bossche, Principal Investigator — University Hospital, Ghent
Locations (1):
- Vakgroep Revalidatiewetenschappen UZ Gent, 1B3, Ghent, Oost-Vlaanderen, Belgium

REFERENCES:
- [Derived] Pringels L, Pieters D, VAN DEN Berghe S, Witvrouw E, Burssens A, Vanden Bossche L, Wezenbeek E. Loading Speed and Intensity in Eccentric Calf Training Impact Acute Changes in Achilles Tendon Thickness and Stiffness: A Randomized Crossover Trial. Med Sci Sports Exerc. 2025 May 1;57(5):895-903. doi: 10.1249/MSS.0000000000003638. Epub 2024 Dec 30. PMID 39787521